CLINICAL TRIAL: NCT01372813
Title: A Phase II Study of ZD6474 (Vandetanib) in Subjects With Advanced Clear Cell Renal Carcinoma
Brief Title: Vandetanib to Treat Advanced Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated for insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, W. Marston Linehan, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080039; 08-C-0039; NCT00608114 (obsolete NCT alias)
Record Dates: First submitted 2011-06-11; First posted 2011-06-14 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Clear Cell Renal Carcinoma
Keywords: Advanced Clear Cell Renal Cell Carcinoma; Cancer; Renal; Renal Cell Carcinoma; Kidney Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Renal Cell; Kidney Neoplasms | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clear Cell Renal Carcinoma (Other): Clear cell renal cancer is a highly vascular tumor characterized by mutations in the von Hippel-Lindau (VHL) gene in the majority of patients, an alteration that leads to overexpression vascular endothelial growth factor (VEGF) as well as other genes such as transforming growth factor-alpha, platelet derived growth factor and glucose transporter 1. Patients received ZD6474 300 mg/day by mouth daily on days 1-28.
  Interventions: Drug: vandetanib

INTERVENTIONS:
Drug: vandetanib — Daily dose 300mg/day by mouth, 28 day cycle
  Other Names: ZD6474

SUMMARY:
Background:

* One way tumors are able to grow is by forming new blood vessels that supply it with nutrients and oxygen.
* Vandetanib (ZD6474) is an experimental drug that blocks certain proteins on the surface of tumor and blood vessel cells that are involved with the formation of new blood vessels.
* Blocking these proteins may prevent the tumor cells or blood vessels from continuing to grow.

Objectives:

* To determine whether vandetanib can cause tumors to shrink or stabilize in patients with advanced kidney cancer.
* To determine how vandetanib may work in people with kidney cancer and to develop tests that may be helpful in studying kidney cancer.

Eligibility:

-Patients 18 years of age or older with advanced clear cell kidney cancer whose disease has worsened after treatment with one or more of the following drugs: sunitinib, sorafenib, interleukin-2 and temsirolimus; or patients who have had to stop treatment with these drugs due to unacceptable side effects; or patients who are unable to receive standard treatment.

Design:

* Patients take a vandetanib pill once a day in 28-day cycles.
* Patients are followed in the clinic every 2 weeks during the first month of treatment and then every 4 weeks for a physical examination, blood and urine tests, electrocardiogram and a review of any drug side effects.
* Patients have imaging scans (computed tomography (CT) or magnetic resonance imaging (MRI)) about every 8 weeks to monitor tumor growth. MRI scans are also done to look at tumor blood flow when treatment begins, 24 hours after the first dose of treatment, and again about 4 and 8 weeks after starting treatment
* Optional tumor biopsies (surgical removal of a sample of tumor tissue) may be done before starting vandetanib treatment and after 4 weeks of treatment to look for drug effects on the tumor.

DETAILED DESCRIPTION:
Background:

* von Hippel-Lindau (VHL) inactivation by mutation or promoter hypermethylation is seen in a high proportion of sporadic clear cell renal cancers.
* Inactivation of VHL leads to accumulation of proteins targeted for degradation through the ubiquitin pathway, which includes a group of transcriptionally active proteins called the hypoxia inducible factors (HIF), whose alpha subunits undergo degradation in a VHL-dependent fashion.
* Accumulation of HIFs results in overexpression of several genes including vascular endothelial growth factor (VEGF), glucose transporter 1 (GLUT-1), transforming growth factor (TGF-a), platelet derived growth factor (PDGF), and erythropoietin, which are believed to play a role in tumorigenesis, tumor progression and metastasis.
* Kinase insert domain-containing receptor/vascular endothelial growth factor receptor 2 (kinase insert domain receptor (KDR)/vascular endothelial growth factor 2 (VEGFR2)) is an endothelial cell receptor for vascular endothelial growth factor (VEGF) and plays a crucial role in mediating tumor angiogenesis, while EGFR (a receptor for TGF-a and epidermal growth factor (EGF) is believed to mediate tumor growth and proliferation.
* ZD6474 is an orally administered receptor tyrosine kinase inhibitor with activity against the KDR/VEGFR2 and the epidermal growth factor receptor (EGFR).

Objective:

Primary Objective

-To evaluate the efficacy (overall response rate) of single agent ZD6474 in advanced clear cell renal cell carcinoma (RCC).

Secondary Objectives

* To evaluate progression free survival in patients treated with ZD6474.
* To study the safety and tolerability of ZD6474.
* To evaluate the correlation between VHL mutational status and response to ZD6474.
* To investigate the effect of ZD6474 on circulating endothelial cells and endothelial progenitor cells and to explore the utility of these markers as surrogates of angiogenesis inhibition.
* To investigate the effect of ZD6474 on potential biomarkers of angiogenesis in plasma such as VEGF and soluble VEGFR2.
* To study the effect of ZD6474 treatment on tumor vascular flow and permeability using dynamic contrast enhanced magnetic resonance imaging.
* To investigate the effect of ZD6474 on EGFR and VEGFR mediated signaling using tumor biopsy tissue (when available).

Eligibility:

* Adults with measurable advanced clear cell renal carcinoma
* Patients must have received no more than three prior systemic therapies (no more than two agents known to inhibit VEGF or VEGFR) and must have either progressed on or be unable to receive 1) Sunitinib or sorafenib, and 2) High dose interleukin-2 (IL-2).

Design:

* Single agent ZD6474 administered daily at a dose of 300mg/day.
* Patients will be evaluated for response every 8 weeks using Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* The study is based on an open label Simon two-stage optimal phase II design and will accrue a maximum of 37 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must meet all the following criteria to be eligible for study enrolment:

Histologically confirmed clear cell renal cell carcinoma (to be confirmed at the Dept. of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI)).

Patients must have advanced disease (metastatic or unresectable) disease.

Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral CT scan.

See section 6.2 for the evaluation of measurable disease.

Prior therapy:

1. All patients must have either received prior sunitinib or sorafenib (discontinued for disease progression or unacceptable toxicity) or be unable to receive these agents. Patients who have discontinued sunitinib or sorafenib for life threatening toxicities that are also known to occur with vandetanib (such as skin, GI toxicities, bowel perforation etc.) will not be eligible.
2. All patients must have failed high dose IL-2, be ineligible to receive this agent or decline this therapy.

   Age greater than or equal to 18 years.

   Life expectancy greater than 3 months.

   Performance status Eastern Cooperative Oncology Group (ECOG) 0-2.

   Patients must have normal organ and marrow function as defined below: white blood cell (WBC) count greater than or equal to 3,000/microL, absolute neutrophil count greater than or equal to 1,500/microL, platelet count greater than or equal to 100,000/microL, serum creatinine less than or equal to 1.5 times upper limit of reference range or measured 24 hr. creatinine clearance greater than or equal to 50 ml/min, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times upper limit of reference range, total bilirubin less than 1.5 times upper limit of reference range (less than 3 times upper limit of reference range in patients with Gilbert's disease), alkaline phosphatase less than or equal to 2.5 times upper limit of reference range (or less than or equal to 5 times upper limit of reference range if considered to be related to liver metastases by the principal investigator (PI))

   Recovery from acute toxicity of prior treatment for RCC (to less than or equal to grade 1 Common Terminology Criteria for Adverse Events (CTCAE) v3.0).

   At least 4 weeks from completion of major surgery and a healed surgical incision.

   Negative pregnancy test in female patients of childbearing potential within 7 days of enrollment.

   Ability to understand and the willingness to sign a written informed consent document.

   EXCLUSION CRITERIA:

   Prior malignancy of other histology, with the exception of cervical carcinoma in situ or adequately treated basal or squamous cell carcinoma of the skin, or any other malignancy for which the patient has not required active treatment for more than three years.

   Patients with VHL disease will be excluded from this study.

   Patients may not be receiving any other investigational agents or have received treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.

   Patients with known brain metastases (except when adequately treated greater than or equal to 6 months before enrollment with no evidence of recurrence).

   Use of 5HT-3 antagonists because of the potential effect on corrected Q wave, T wave (QTc) interval.

   Any concurrent medication that may cause QTc prolongation or induce Torsades de Pointes (Appendix C).

   Drugs listed in Appendix C, Table 2, that in the investigator's opinion cannot be discontinued, are allowed, but must be monitored closely.

   Clinically significant cardiac event (including symptomatic heart failure, myocardial infarction or angina) within 3 months of entry or presence of any cardiac disease that in the opinion of the Principal Investigator increases the risk of ventricular arrhythmia.

   Patients with a history a major cardiac event more than 3 months prior to enrolment will be evaluated by a cardiologist to assess cardiac status and potential for increased risk with ZD6474 therapy.

   History of clinically significant arrhythmia [including multifocal premature ventricular contraction (PVC), bigeminy, trigeminy, ventricular tachycardia] that is symptomatic or requires treatment (CTCAE grade 3) or symptomatic/ asymptomatic sustained ventricular tachycardia.

   Uncontrolled atrial fibrillation. Atrial fibrillation controlled on medication is not excluded.

   Presence of Left bundle branch block.

   Previous history of QTc prolongation while taking other medications that required discontinuation of that medication.

   Congenital long QT syndrome or first degree relative with unexplained sudden death under the age of 40 years.

   QTc with Bazett's correction that is unmeasurable, or greater than or equal to 480 msec on screening ECG.

   If a patient has QTc greater than or equal to 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart).

   The average QTc from the three screening electrocardiograms (ECGs) must be less than 480 msec in order for the patient to be eligible for the study).

   Patients who are receiving a drug that has a risk of QTc prolongation (see Appendix C, Group/Table 2) are excluded if QTc is greater than or equal to 460 msec.

   Potassium concentration less than 4.0 mEq/L, calcium (ionized calcium or adjusted for albumin), or magnesium concentrations outside normal limits despite optimal supplementation/correction.

   Left ventricular ejection fraction less than 45 percent measured by multiple gated acquisition scan (MUGA) or echocardiogram (ECHO).

   Hypertension not controlled by medical therapy (systolic blood pressure greater than 150 mmHg or diastolic blood pressure greater than 100 mmHg).

   Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

   Patient known to be human immunodeficiency virus (HIV)-positive and requiring antiretroviral therapy.

   Currently active diarrhea that may affect the ability of the patient to absorb ZD6474 or tolerate further diarrhea.

   Pregnant women are excluded from this study because ZD6474 is an anti-angiogenic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ZD6474, breastfeeding should be discontinued if the mother is treated with ZD6474.

   Any known hypersensitivity to ZD 6474 or other excipients of ZD6474.

   Concomitant medications that are potent inducers of cytochrome P450 3A4 (CYP3A4) function, such as rifampin, rifabutin, phenytoin, carbamazepine, barbiturates such as phenobarbital, or St. John's Wort.

   Inclusion of Women and Minorities:

   Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Marston Linehan, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Zambrano NR, Lubensky IA, Merino MJ, Linehan WM, Walther MM. Histopathology and molecular genetics of renal tumors toward unification of a classification system. J Urol. 1999 Oct;162(4):1246-58. PMID 10492174
- [Background] Chow WH, Devesa SS, Warren JL, Fraumeni JF Jr. Rising incidence of renal cell cancer in the United States. JAMA. 1999 May 5;281(17):1628-31. doi: 10.1001/jama.281.17.1628. PMID 10235157
- [Background] Phillips JL, Pavlovich CP, Walther M, Ried T, Linehan WM. The genetic basis of renal epithelial tumors: advances in research and its impact on prognosis and therapy. Curr Opin Urol. 2001 Sep;11(5):463-9. doi: 10.1097/00042307-200109000-00003. PMID 11493766
- See also: Medline — http://www.nlm.nih.gov/medlineplus
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: US FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial only accrued 3 participants.
Groups:
- Clear Cell Renal Carcinoma Patients: Clear cell renal cancer is a highly vascular tumor characterized by mutations in the von Hippel-Lindau (VHL) gene in the majority of patients, an alteration that leads to overexpression vascular endothelial growth factor (VEGF) as well as other genes such as transforming growth factor-alpha, platelet derived growth factor and glucose transporter 1. Patients received ZD6474 300 mg/day by mouth daily on days 1-28.
Period: Overall Study
Arm/Group | Clear Cell Renal Carcinoma Patients
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (5.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Response (Partial Response (PR) + Clinical Response (CR))
Description: Clinical response is the best response recorded from the start of treatment until disease progression. Clinical response is assessed by the Response Evaluation in Solid Tumors (RECIST) criteria. A partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as a reference the baseline sum LD. A complete response (CR) is the disappearance of all target lesions.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Effect of Vandetanib on Plasma Biomarkers-vascular Endothelial Growth Factor (VEGF), Vascular Endothelial Growth Factor 2 (VEGFR2)
Description: Plasma VEGFR and VEGFR2 would have been measured using the (enzyme-linked immunosorbent assay)ELISA at baseline and specified timepoints following initiation of therapy.
Time Frame: 12 months
Population: Not enough samples for meaningful analysis.
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Circulating Endothelial Progenitor Cells (CEP) Per 10^6 Mononuclear Cells or Per Microliter of Peripheral Blood Analyzed in Samples Taken Before and After Treatment
Description: CEP cell concentrations are calculated as a percentage of the total number of mononuclear cells or as the number of cells/microliter of whole blood after an evaluation of a minimum of 10^5 cellular events, and preferably 10^6 cellular events.
Time Frame: 12 months
Population: Not enough samples for meaningful analysis.
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival as Defined by the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Progression free survival is defined as the time from initiation of treatment to either progression or death.
  RECIST evaluates tumor response. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria. For detailed information about RECIST, see the protocol Link module.
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 3
Days | 55 [51 to 111]

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 11.5 months
Measure: Number; unit: Participants
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 3
Participants | 3

6. Secondary Outcome: Number of Circulating Endothelial Cells (CEC) Per 10^6 Mononuclear Cells or Per Microliter of Peripheral Blood Analyzed in Samples Taken Before and After Treatment
Description: CEC cell concentrations are calculated as a percentage of the total number of mononuclear cells or as the number of cells/microliter of whole blood after an evaluation of a minimum of 10^5 cellular events, and preferably 10^6 cellular events.
Time Frame: 12 months
Population: Not enough samples for meaningful analysis.
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Vandetanib (ZD6474) Effects on Tumor Vascular Flow and Permeability Using Dynamic Contrast Enhanced Magnetic Resonance Imaging (DCE-MRI)
Description: Flow dynamics within specific tumor sites will be evaluated based on the results of the DCE-MRI obtained first without contrast enhancement and then after contrast enhancement. The parameter to be measured is the forward contrast transfer rate (Ktrans), the reverse contrast transfer rate (Kep), and/or the extravascular extracellular space volume fraction (Ve). Flow dynamics are a measure of blood flow changes in the tumor and are determined using the parameters previously defined (Ktrans, Kep, etc.).
Time Frame: 12 months
Measure: Number; unit: Participants with changes
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 2
Participants with changes | 0

8. Secondary Outcome: Tumor Tissue Used to Evaluate Von Hippel-Lindau (VHL) Status and/or Components of the Vascular Endothelial Growth Factor (VEGF)/Epidermal Growth Factor Receptor (EGFR) Pathway
Description: Components of the VEGF and EGFR pathways were to be evaluated using Western blot analysis at baseline and specified timepoints following initiation of therapy when tumor tissue was available.
Time Frame: 12 months
Population: Not enough samples for meaningful analysis.
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 0

9. Secondary Outcome: The Effects of ZD6474 (Vandetanib) on Tumor Microvessel Density
Description: Tumor tissue sections were to be stained with hematoxylin and eosin (H and E) and endothelial cell markers at baseline and specified timepoints following initiation of therapy (when tumor tissue was available)
Time Frame: 12 months
Population: Not enough samples for meaningful analysis.
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 0

10. Secondary Outcome: Evaluate The Correlation Between Von Hippel-Lindau (VHL) Mutational Status and Response to ZD6474 (Vandetanib)
Description: If an adequate number of responses were seen, the relation of these responses to the presence/absence of inactivating VHL mutations in tumor tissue would have been assessed.
Time Frame: 12 months
Population: Not enough samples for meaningful analysis.
Arm/Group | Clear Cell Renal Carcinoma Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 11.5 months
Arm/Group | Clear Cell Renal Carcinoma Patients
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clear Cell Renal Carcinoma Patients (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clear Cell Renal Carcinoma Patients (N=3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Bicarbonate, serum-low (Investigations) | 1 (1)
Creatinine (Investigations) | 1 (1)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Neurology - Other (Specify, lightheadedness) (Nervous system disorders) | 1 (1)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1) — Neck and shoulder
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Prolonged QTc interval (Investigations) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was designed to accrue up to 37 patients but only 3 were enrolled. Study was terminated due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No